CLINICAL TRIAL: NCT01946308
Title: Sleep Organization in Premature Infants With Feeding Difficulties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CHMC 2011-1456
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2013-09

CONDITIONS: Premature Infant Sleep
Keywords: sleep; sleep efficiency; active sleep; quiet sleep; arousals; premature infant; conformational positioning; mattress; feeding difficulty; neonatal intensive care unit; sleep state; behavioral observation; stress behavior; self-regulatory behavior; surgery; gastrointestinal
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- conformational positioner & mattress (Experimental): conformational positioner & mattress, five hours on each
  Interventions: Other: Conformational positioning system

INTERVENTIONS:
Other: Conformational positioning system — The conformational positioning system will be compared to the standard infant crib mattress.
  Other Names: therapeutic positioner; fluidized bed positioner

SUMMARY:
Babies born too soon, premature babies, can have complications following birth because their systems are immature. Hospitals help prevent deformities and delays in motor development by using therapeutic positioning to provide containment as they would experience in the womb. They also often have trouble eating. They have discomfort, are irritable, refuse to eat and cry because their digestive system is immature. The neonatal intensive unit can create stress and disrupt their sleep. Going from active to deep sleep is essential for infant brain development, learning and memory formation. Their sleep states early in life predict their developmental outcome. The purpose is to determine whether a conformational positioning system, one that can mold to the baby and contain him or her, will allow more time asleep in premature infants with feeding problems compared to the standard crib mattress. We hypothesize that the number of total sleep time will be longer and the number of arousals out of sleep lower when they are sleeping on the conformational positioning system compared to the mattress.

DETAILED DESCRIPTION:
Premature infants are at risk for complications due to the immaturity of motor, gastrointestinal, respiratory, cutaneous and behavioral systems. Therapeutic positioning is routinely used to provide containment, maintain a flexed position and prevent skeletal deformities and delays in motor development. Premature infants have feeding difficulties and frequently experience gastroesophageal reflux, discomfort, refusal to feed, irritability, and crying. The neonatal intensive care environment can create stress and disrupts sleep-wake cycles and self-regulatory behaviors. Cycling from active to deep sleep states is required for neurosensory processing, learning, memory formation and brain plasticity. Sleep and waking states for premature infants are predictive of neurodevelopmental outcomes. The purpose of the study is to determine whether the use of conformational positioning will be associated with greater total sleep time in premature infants with a history feeding difficulty compared to positioning on a mattress alone. We hypothesize that the number of arousals and total sleep time will be affected by the support surface. Specifically, the number of arousals will be lower and total sleep time will be greater for infants when they are on a conformational positioning (CP) device compared to when they are on the standard positioning system (mattress) (SP). The use of CP will reduce the number of arousals, increase the total sleep time, and bring about behavioral states that are conducive to regulation of attention, state and motor response relative to SP.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of < 37 weeks
* Feeding difficulty due to prematurity or a medical condition
* Not taking sedative medications for 24 hours before sleep study
* Post-surgery
* Sufficiently medically stable to undergo procedures

Exclusion Criteria:

* Gestational age equal to or greater than 37 weeks
* Clinical apnea
* Require mechanical ventilatory support
* Received sedative medications 24 hours before sleep study
* Brain injury or neurological condition that limits movement
* Orthopedic conditions requiring fixed positioning
* Arthrogryposis
* Osteogenesis imperfecta
* Medically unstable such that procedures cannot be tolerated

Ages: 26 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Sleep organization defined as efficiency, active sleep time, quiet sleep time, number of arousals, measured by polysomnography | Overnight, 10.5 hour standard EEG sleep study
  Standard polysomnography electrodes are applied to the subject in the evening and the subject is placed on either the standard mattress or the conformational positioning system (assigned at random) for the first 5 hours. The subject is then moved onto the second treatment for the remainder of the study. EEG measures are recorded continuously over the entire period. The EEG data are assessed by trained sleep study physicians and clinical staff.

SECONDARY OUTCOMES:
Sleep state by behavioral observation | Two 30-minute periods, one on each treatment, during the EEG sleep study
  Nurses trained in the techniques of premature infant behavioral state determination will observe the infant for two 30-minute periods while the EEG sleep study is being conducted. One nurse will observe when the subject is on the standard mattress and the other will observe when the subject is on the conformational positioning system. They will record specific behaviors observed in 2-minute intervals during the 30-minute period.

OTHER OUTCOMES:
Impact of prior surgery on sleep organization | Overnight, 10-hour sleep study
  Standard polysomnography electrodes are applied to the subject in the evening and the subject is placed on either the standard mattress or the conformational positioning system (assigned at random) for the first 5 hours. The subject is then moved onto the second treatment for the remainder of the study. EEG measures are recorded continuously over the entire period. The EEG data are assessed by trained sleep study physicians and clinical staff. The sleep organization and behaviorally observed sleep state will be compared for the subjects grouped as having had surgery prior to the study or not having had surgery to ascertain the impact of surgery while controlling for the treatment effects.

CONTACTS AND LOCATIONS:
Overall Officials: Marty O Visscher, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Visscher MO, Lacina L, Casper T, Dixon M, Harmeyer J, Haberman B, Alberts J, Simakajornboon N. Conformational positioning improves sleep in premature infants with feeding difficulties. J Pediatr. 2015 Jan;166(1):44-8. doi: 10.1016/j.jpeds.2014.09.012. Epub 2014 Oct 12. PMID 25311708